CLINICAL TRIAL: NCT03129451
Title: The Microbiome in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Ashok Sriram, Principal Investigator, Corewell Health West
Other Study IDs: 2016-313
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Tremor-dominant: Tremor-dominant Parkinson's disease
  Interventions: Diagnostic Test: Microbiome specimens in stool
- Akinetic-Rigid: Akinetic-Rigid type Parkinson's disease
  Interventions: Diagnostic Test: Microbiome specimens in stool
- Multiple systems atrophy: Multiple systems atrophy PD
  Interventions: Diagnostic Test: Microbiome specimens in stool
- Levodopa-naïve: Levodopa-naïve Parkinson's disease
  Interventions: Diagnostic Test: Microbiome specimens in stool
- Tremor-dominant / app: Tremor-dominant Parkinson's disease with an appendectomy
  Interventions: Diagnostic Test: Microbiome specimens in stool
- Akinetic-Rigid / app: Akinetic-Rigid Parkinson's disease with an appendectomy
  Interventions: Diagnostic Test: Microbiome specimens in stool
- Levodopa-naïve w/app: Levodopa-naïve Parkinson's disease with an appendectomy
  Interventions: Diagnostic Test: Microbiome specimens in stool

INTERVENTIONS:
Diagnostic Test: Microbiome specimens in stool — Analyzing Microbiome specimens in stool

SUMMARY:
To investigate the dynamic relationship between the intestinal microbiota and Inflammation in subjects with Parkinson's disease.

DETAILED DESCRIPTION:
To investigate the dynamic relationship between the intestinal microbiota and Inflammation in subjects with Parkinson's disease. The current study examines the differential microbiome of the gut in subjects with parkinsonism. The current study determines whether certain Parkinson's subtypes are prone to pro-inflammatory microbiomes. This study also explores whether the intestinal microbiome in post-appendectomy Parkinson's subjects is modified as appendix has a role in regulating intestinal microbiome. The current study will examine whether microbiome changes influence inflammatory markers in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Parkinson's disease (including multiple system atrophy). Males and females are eligible for the study. Appendectomized cohort must have had their appendectomy at least 20 years before Parkinson's disease onset

Exclusion Criteria:

* 1. Body Mass Index greater than or equal to 35 or less than or equal to 18. 2. Vital signs outside of acceptable range at Screening Visit, i.e., blood pressure >160/100, oral temperature >100°F, pulse >100.

  3. Use of any of the following drugs within the last 6 months:
  * systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral);
  * cytokines;
  * methotrexate or immunosuppressive cytotoxic agents;
  * large doses of commercial probiotics consumed (greater than or equal to 108 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.

    4. Acute viral/bacterial infection disease at the time of sampling (defer sampling until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever.

    5. Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.

    6. Recent history of chronic alcohol consumption defined as more than five 1.5- ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day.

    7. Positive test for HIV, HBV or HCV. 8. Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection.

    9. Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.

    10. History of active uncontrolled gastrointestinal disorders or diseases including:
  * inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis;
  * irritable bowel syndrome (IBS) (moderate-severe);
  * persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated); 11. Female who is pregnant or lactating. 12. Atypical or secondary Parkinson's disease 13. Adults that are unable to consent, individuals that are not yet adults and prisoners are not eligible for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will examine individuals who are current patients of a Spectrum Health Movement Disorder physician with: 1) Tremor-dominant Parkinson's disease, 2) Akinetic-Rigid type Parkinson's disease, 3) Multiple systems atrophy (MSA-P), 4) Levodopa-naïve Parkinson's disease, 5) Tremor-dominant Parkinson's disease with an appendectomy, 6) Akinetic-Rigid Parkinson's disease with an appendectomy, 7) Levodopa-naïve Parkinson's disease with an appendectomy
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
The current study determines whether certain Parkinson's subtypes are prone to pro-inflammatory microbiomes. | 3 years
  Differences in microbiome abundance will be detected using a Kruskal-Wallis' test generating a Benjamini-Hochberg false discovery rate (FDR)-corrected P value (<0.05 for significance). For the microbiome analysis, in silico community functional predictions will be performed using PICRUSt (Phylogenetic Investigation of Communities by Reconstruction of Unobserved States) and significant differences in Kyoto Encyclopedia of Genes and Genomes (KEGG) ortholog (KO) abundances between groups will be identified (FDR-corrected P value <0.05 for significance). Putative "proinflammatory" and "anti-inflammatory" bacteria taxa will be classified based on previous reports (and the references therein) (see Keshavarzian et al., 2015). Differences in inflammatory metabolite abundance will be detected using a Kruskal-Wallis' test generating a Benjamini-Hochberg false discovery rate (FDR)-corrected P value (0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Sriram, MD, MS, Principal Investigator — Spectrum Health Medical Group
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No